CLINICAL TRIAL: NCT06423144
Title: A Retrospective Study Comparing Interventional Therapy (TACE/HAIC) Combined With PD-1/PD-L1 Inhibitors and Anti-angiogenic Agents Versus PD-1/PD-L1 Inhibitors and Anti-angiogenic Agents Alone in the First-line Treatment of Intermediate and Advanced Hepatocellular Carcinoma Beyond up to Seven
Brief Title: PD-1/PD-L1 Inhibitors and Anti-angiogenic Therapy Combined With/Without TACE/HAIC in Patients With BCLC B/C Hepatocellular Carcinoma Beyond Up-to-7
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Lan Zhang, Chief physician, Shanghai Zhongshan Hospital
Other Study IDs: ZL-2024-06
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Angiogenesis Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group LS: Logical therapy combined with systemic therapy
  Interventions: Procedure: TACE/HAIC; Drug: PD-1/PD-L1 inhibits and anti-angiogenic agents
- Group S: Systemic therapy alone（PD-1/PD-L1 inhibits and anti-angiogenic agents）
  Interventions: Drug: PD-1/PD-L1 inhibits and anti-angiogenic agents

INTERVENTIONS:
Procedure: TACE/HAIC — TACE/HAIC were performed within 1 month prior/after the first PD-1/PD-L 1 inhibitor/antiangiogenic drug treatment;
  Groups: Group LS
Drug: PD-1/PD-L1 inhibits and anti-angiogenic agents — Agents were administrated based on the instructions recommended

SUMMARY:
This is a retrospective study that retrospectively included patients with intermediate and advanced HCC beyond up to seven who received first-line treatment with PD-1/PD-L1 inhibitors and anti-angiogenic agents combined with/without TACE/HAIC from January 01, 2019 to December 31, 2023 in the Department of Hepatic Oncology and Department of Liver Cancer Surgery, Zhongshan Hospital, Fudan University.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with advanced hepatocarcinoma (HCC), confirmed histologically or clinically.
* Patients with Barcelona (BCLC) stage B and C beyond up to seven;
* Have not received any prior systemic therapy for HCC (including: chemotherapy, molecular targeted therapy, immunotherapy);
* Receiving only post-marketing PD-1/PD-L1 inhibitors in combination with anti-angiogenic agents (including, but not limited to, drugs containing hepatocellular carcinoma indications);

  *The interval between the first use of PD-1/PD-L 1 inhibitors and the use of anti-angiogenic drugs is ≤ 1 week
* TACE was performed within 1 month prior/after the first PD-1/PD-L 1 inhibitor/antiangiogenic drug treatment;
* TACE treatment followed by at least 1 cycle of combination therapy, including: cTACE and DEB-TACE;
* There is at least 1 measurable lesion in the liver according to RECIST v1.1 criteria

Exclusion Criteria:

* Cholangiocellular carcinoma, mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, or hepatic fibrous laminar carcinoma that has been pathologically/histologically confirmed;
* Patients who do not meet the above definition of combination therapy;
* Patients had malignant tumors other than HCC within 5 years prior to enrollment (except cured limited tumors, including cervical carcinoma in situ, basal cell carcinoma of the skin, and prostate carcinoma in situ)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate and advanced hepatocellular carcinoma beyond up to seven
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 48 months
  The time from the beginning of treatment to the time of tumor progression or death from any cause (according to mRECIST and RECIST v1.1)
ORR | Up to 48 months
  The percentage of patients who have best overall response of complete response (CR) or partial response (PR) according to mRECIST and RECIST v1.1

SECONDARY OUTCOMES:
OS | Up to 48 months
  OS was defined as the interval from the date of the initial administration of any drug/procedure to death from any cause.
Safety | Up to 48 months
  Safety was defined the incidence and severity of adverse events (AEs) and serious adverse events (SAEs). The severity of AEs were evaluated based on the National Cancer Institute Common Terminology Criteria for Adverse Events version (NCI-CTCAE) v5.0.

IPD SHARING:
Plan to Share IPD: Undecided